CLINICAL TRIAL: NCT03639038
Title: Reagent Evaluation Plan: Tuberculosis Diagnosis by Flow Cytometry (Project Orion)
Brief Title: Tuberculosis Diagnosis by Flow Cytometry
Status: Withdrawn | Type: Observational
Why Stopped: PI retired, study never opened.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Stewart Reid, co-investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300001699
Record Dates: First submitted 2018-08-14; First posted 2018-08-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Blood Assay Phase - 1: TB Positive / HIV Positive: 65 participants
- Blood Assay Phase - 2: TB positive / HIV Negative: 65 participants
- Blood Assay Phase - 3: TB positive and negative Paediatric: 30 participants
- Blood Assay Phase - 4: TB Negative/HIV positive: 50 participants
- Blood Assay Phase - 5: Healthy controls: 30 participants
- Sputum Collection Phase - 1: TB Positive: Xpert Rif sensitive: 100 participants
- Sputum Collection Phase - 2: TB Positive: Xpert Rif resistant: 20
- Sputum Collection Phase - 3: TB Negative: Other chest: unknown number
- Sputum Collection Phase - 4: TB Negative: Smear negative/Xpert negative: 20

SUMMARY:
Tuberculosis and HIV continue to be major public health problems in resource constrained settings like Zambia. Zambia is among the top 30 highest burden countries globally. The major drivers of TB in the Africa region is the HIV epidemic. Inadequate TB diagnostic tools with failure to make a timely diagnosis and start appropriate treatment are the major impediments to TB control in Zambia and globally.

DETAILED DESCRIPTION:
Project Orion is focused on utilizing Flow Cytometry Technology to screen and diagnose tuberculosis. There are two assays being tested under this Project:

1. Activated TB assay for differentiation of latent and active TB infection using blood samples and
2. Direct TB assay (DTA) for rapid detection and DST of Mycobacterium tuberculosis (Mtb) using sputum specimens.)

ELIGIBILITY:
Inclusion Criteria:

* Presumptive TB patients (patients recommended for tuberculosis diagnostic testing and not on ATT)
* Patients with multi-drug resistant TB (MDR-TB)
* Paediatric patients (< 15 years old)
* Patients suspected of extra-pulmonary tuberculosis
* Patients with TB/HIV co-infection

Exclusion Criteria:

* Unable/unwilling to sign Informed consent

Ages: 5 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be selected on a first come, first serve basis at TB clinics in MOH District clinics in Lusaka. The participants will include both confirmed TB patients as well as presumptive TB patients. All participants should not have started anti-TB treatment (ATT) prior to enrollment or be less than five days from treatment start.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-09-30 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
ATB assay for differentiation of latent and active TB infection using Blood samples | The duration of this project is 9 months.
  To evaluate the clinical utility of the test reagent(s) compared to diagnostic gold Standard: Culture and Xpert MTB/Rif along with clinical (empiric) diagnosis
DTB assay for rapid detection and drug sensitivity testing of Mtb using sputum specimens | The duration of this project is 9 months.
  To evaluate the clinical utility of the test reagent(s) compared to diagnostic gold Standard: Culture and Xpert MTB/Rif along with clinical (empiric) diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Monde Muyoyeta, MD, PhD, Principal Investigator — Center for Infectious Disease Research in Zambia
Locations (1):
- Center for Infectious Disease Research in Zambia (CIDRZ), Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No